CLINICAL TRIAL: NCT05116358
Title: Phase II Study - Trial of a Phototherapy Light Device to Improve Sleep Health
Acronym: PHOTONS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: CeraZ LLC (Unknown)
Responsible Party: Principal Investigator, MICHAEL A GRANDNER, Assistant Professor of Psychiatry, Psychology, and Medicine; Director, Sleep & Health Research Program, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012256803
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Phase II Interventional (Clinical Trial) Determine whether use of the light therapy device (versus sham device) results in changes to self-reported sleep quality, self-reported sleep continuity, objectively-estimated sleep continuity, and objectively-estimated sleep architecture. Additionally, to determine whether use of the light therapy device (versus placebo device) results in improvements in mood and daytime functioning .and induce improvements in mood, stress, morning energy levels, perceived daytime functioning, and fatigue levels.
Who Masked: Participant
Masking Description: Phase II - Masked (Sham Controlled) Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): An active phototherapy device
  Interventions: Device: Phototherapy device
- Sham (Placebo) (Sham Comparator): An inactive device
  Interventions: Device: Phototherapy device

INTERVENTIONS:
Device: Phototherapy device — The active phototherapy device will emit light

SUMMARY:
There are few devices currently on the market claiming to improve sleep. This study will investigate the efficacy of phototherapy on improving sleep, in the form of a wearable neck device used at night.

DETAILED DESCRIPTION:
This study will investigate the efficacy of phototherapy on improving sleep, in the form of a wearable neck device used at night. Phototherapy has been shown to improve chronic pain, cerebral blood flow, neurological function, and capillary growth in skeletal muscle. A device worn at night may improve sleep onset, total sleep time, or modify sleep architecture. Improved cardiovascular function may facilitate a decrease in core body temperature needed for sleep onset. Relaxation from direct heat may help to decrease cortisol levels, thus reducing the number of night-time arousals. It may also decrease circulating levels of norepinephrine (NE), one of the main neurotransmitters involved in arousal. The aim of this study is to evaluate if the device worn leads to greater next-day wellbeing and cognitive function as a result of increased slow-wave activity.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 60 years old
2. Able to read and write fluently in English
3. Access to a mobile device for video calls, online questionnaires, syncing devices, and communication with study staff
4. Access to a residential mailing address for shipping study materials
5. Exhibit a score of >8 on the Insomnia Severity Index
6. Self-report that they have a problem with their sleep that they wish to improve

Exclusion Criteria:

1. Have a moderate to severe current sleep disorder
2. Have a current psychiatric disorder
3. Are taking medication that would interfere with sleep, including beta blockers, antidepressants, antianxiety medications, hypnotics, or stimulants
4. Have a medical condition that would interfere with their ability to complete all study procedures or would render measurements invalid (e.g., some autoimmune conditions, cardiac conditions, endocrine conditions, or chronic pain conditions)
5. Exhibit a regular sleep schedule, where bed and wake times are kept within a 2-hour window 7 days per week
6. Exhibit a regular sleep schedule during the night, beginning no earlier than 9pm and ending no later than 10am
7. Have not engaged in shift work for the past month, and will refrain from shift work during the study
8. Are unable to restrict alcohol consumption to no more than 2 drinks within 4 hours of sleep
9. Are unable to restrict caffeine use to no coffee or caffeinated beverages after 12pm during the study
10. Regularly smoke or use other tobacco products
11. Regularly use cannabis-derived medicinal products
12. Are pregnant
13. Are a full-time caregiver to an individual that requires attending during the evening and night

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in subjective rating of the device across a 3-week intervention | Change in subjective rating of the device from baseline (pre; Day 0) to after 21 days of wearing it (post)
  There will be a subjective rating of the phototherapy device using a series of questions assessing device's effect on sleep and next-day function at the end of the trial.
Change in Insomnia Severity Index (ISI) scores across a 3-week intervention | Change from baseline over the course of the study (after 21 days of wearing the device)
  The ISI is a 7-item insomnia screening tool that is the gold standard for quantifying severity of clinical insomnia symptoms.
Change in objective sleep efficiency across a 3-week intervention | Change from mean baseline period (first two weeks of wear) to post three weeks of wearing the phototherapy device.
  Objective sleep efficiency will be measured with a wearable device (Oura ring) that is worn for the duration of the study and captures sleep and wake data using actigraphy.

SECONDARY OUTCOMES:
Change in mean sleep latency assessed using sleep diaries | Change from mean baseline period (first two weeks of wear) to post three weeks of wearing the phototherapy device.
  Sleep latency, or time taken to fall asleep, will be assessed using morning sleep diaries completed by the participant upon awakening. The mean sleep latency during the baseline period (pre) will be compared to after three weeks of wearing the phototherapy device (post).
Change in Karolinska Sleepiness Scale (KSS) score | Change from before intervention (pre) to post three weeks of wearing the phototherapy device (Day 21)..
  The Karolinska Sleepiness Scale (KSS) measures situational sleepiness on a 9-point scale
Circadian Energy Scale (CIRENS) score | Change from baseline (pre) to post three weeks of wearing the phototherapy device (Day 21).
  CIRENS is a very short and simple chronotype measurement tool based on energy. The CIRENS consists of two introspective questions about the usual energy level (very low, low, moderate, high, or very high, scored 1 to 5) in the morning and in the evening. The difference between energy level scores (-4 to 4) felt by respondents in the evening and morning defines the chronotype score and classification.
Positive and Negative Affect Scales (PANAS) Positive Affect | Change from baseline (pre) to post three weeks of wearing the phototherapy device (Day 21).
  The Positive and Negative Affect Scales are brief screening measures that assess both positive and negative emotional experiences. This scale will allow for separate assessment of impact on positive mood.
Positive and Negative Affect Scales (PANAS) Negative Affect | Change from baseline (pre) to post three weeks of wearing the phototherapy device (Day 21).
  The Positive and Negative Affect Scales are brief screening measures that assess both positive and negative emotional experiences. This scale will allow for separate assessment of impact on negative mood.
Change in Fatigue Severity Scale (FSS) across a three-week intervention | Change from baseline (pre) to post three weeks of wearing the phototherapy device (Day 21).
  Fatigue Severity Scale (FSS) is a well-validated 9-item clinical measure that assesses overall levels of mental and physical fatigue, with answers ranging from 1- "Strongly Disagree" to 7-"Strongly Agree".
Change in Profile of Mood States (POMS) across a three week intervention | Change from baseline (pre) to post three weeks of wearing the phototherapy device (Day 21).
  The Profile of Mood States (POMS) is a psychological rating scale used to assess transient, distinct mood states. The POMS measures six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment. A total score will be evaluated in addition to the individual items.
Change in Wake After Sleep Onset (WASO) assessed using morning sleep diaries over the duration of the study | Change from mean baseline period (first two weeks of wear) to post three weeks of wearing the phototherapy device.
  Wake after sleep onset (WASO), or the number of nocturnal awakenings, will be assessed using morning sleep diaries completed by the participant upon awakening. The mean WASO during the baseline period (pre) will be compared to after three weeks of wearing the phototherapy device (post).
Change in sleep efficiency assessed using morning sleep diaries over the duration of the study | Change from mean baseline period (first two weeks of wear) to post three weeks of wearing the phototherapy device.
  Sleep efficiency, or the amount of time spent asleep during a sleep opportunity, will be assessed using morning sleep diaries completed by the participant upon awakening. The mean sleep efficiency during the baseline period (pre) will be compared to after three weeks of wearing the phototherapy device (post).
Change in total sleep time assessed using morning sleep diaries over the duration of the study | Change from mean baseline period (first two weeks of wear) to post three weeks of wearing the phototherapy device.
  Total sleep time will be assessed using morning sleep diaries completed by the participant upon awakening. The mean total sleep time during the baseline period (pre) will be compared to after three weeks of wearing the phototherapy device (post).
Change in morning refreshed feeling assessed using morning sleep diaries over the duration of the study | Change from mean baseline period (first two weeks of wear) to post three weeks of wearing the phototherapy device.
  Morning refreshed feeling will be assessed using morning sleep diaries completed by the participant upon awakening. The mean refreshed feeling during the baseline period (pre) will be compared to after three weeks of wearing the phototherapy device (post).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kennedy KER, Wills CCA, Holt C, Grandner MA. A randomized, sham-controlled trial of a novel near-infrared phototherapy device on sleep and daytime function. J Clin Sleep Med. 2023 Sep 1;19(9):1669-1675. doi: 10.5664/jcsm.10648. PMID 37141002